CLINICAL TRIAL: NCT04559516
Title: Remote Exercise Program deliVery Using A Mobile Phone Application for Patients With Pulmonary Arterial Hypertension (REVAMP): a Pilot Randomized Trial
Brief Title: Remote Exercise Program Delivery Using a Mobile Application for Pulmonary Arterial Hypertension
Acronym: REVAMP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator moved to different institution.
Sponsor: University of Calgary (Other)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0184
Record Dates: First submitted 2020-09-04; First posted 2020-09-23 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Rehabilitation; Mobile-based home exercise program
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Standard of Care

STUDY DESIGN:
Masking Description: The principal investigator and co-investigator will be unaware of allocation until after the beginning of the exercise program. There will be no blinding after intervention begins, as is typical with studies of exercise intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application-based home exercise intervention (Experimental): The exercise program will be administered over 12 weeks through the Ethica mobile app. Participants will perform exercise sessions at home guided by instructional video accessed via Ethica, six days per week. The program will include a combination of education, endurance, strength, and respiratory muscle training.
  The Ethica mobile app will provide a daily alert and a daily exercise video. There will be background monitoring of step counts and actigraphy will be monitored for one week intervals at baseline, at week six, and at week twelve.
  Interventions: Behavioral: Exercise Intervention
- Standard care (Active Comparator): No supervised exercise session will be performed. Symptoms and quality of life will be monitored in the same manner as the intervention group, and participants will receive the same educational message alerts through the Ethica app as the exercise intervention group.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Exercise Intervention — The Ethica mobile app will provide a daily alert accompanied by a short educational statement about PAH, disease self-management tips, dietary and nutritional advice, goal setting, and a motivational statement to encourage patients.
  Participation with each session will be assessed by a mobile app-embedded survey administered at the end of the day. Patients will be presented with weekly alerts to complete validated patient-reported quality of life questionnaires using the EmPHasis-10 and the Living with Pulmonary Hypertension Questionnaire, as well as the PRAISE self-efficacy score for pulmonary rehabilitation. The app will also ask patients to report their WHO/NYHA functional class every week. Using in-app buttons, participants can log adverse events associated with each exercise session.
  Arms: Mobile application-based home exercise intervention
Behavioral: Standard Care — Participants will be provided usual care administered at the PH clinic at the University of Calgary and no supervised exercise session will be performed.
  Arms: Standard care

SUMMARY:
This study will determine the feasibility of a mobile application-based home exercise rehabilitation program for patients with pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary rehabilitation programs that incorporate exercise training are an important component of optimal medical care for pulmonary arterial hypertension (PAH) and chronic thromboembolic pulmonary hypertension (CTEPH), which improves exercise performance, quality of life, and may even modify disease progression.

To date, no studies have utilized mobile health (mHealth) technology to provide exercise program interventions in the pulmonary hypertension population. Leveraging mobile technology, such as smartphones or tablets, to administer a home-based exercise rehabilitation program could improve patient access, satisfaction, and participation, while providing sustained physiologic benefits and incurring major cost savings compared to inpatient or outpatient-based supervised programs.

This study hypothesis is that a home-based exercise program delivered by a mobile app will be feasible and safe for PAH/CTEPH patients. The secondary outcomes assessed will explore whether there are changes in exercise capacity, health-related quality of life, and right ventricular function, compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.

   Either 2 OR 3
2. Diagnosis of PAH by a right heart catheterization with documented mean pulmonary arterial pressure (mPAP) ≥ 20 mmHg, pulmonary arterial wedge pressure ≤ 15 mmHg and a pulmonary vascular resistance (PVR) > 3 wood units.
3. Diagnosis of CTEPH with mPAP ≥ 20 mmHg, pulmonary arterial wedge pressure ≤ 15 mmHg and a pulmonary vascular resistance (PVR) > 3 wood units. Evidence of thromboembolic occlusion of the pulmonary arterial system. The patient must be deemed inoperable for, or have persistent pulmonary hypertension after, thromboendarterectomy.
4. Must own a mobile smart phone or tablet and have internet access at home.
5. Stable doses of PAH medications for ≥3 months. Changes to diuretic doses or anticoagulation within 3 months are permitted.

Exclusion Criteria:

1. High-risk PAH, defined as REVEAL 2.0 score ≥9 or high-risk according to the 2015 European Society of Cardiology/European Respiratory Society (ESC/ERS) guidelines table.
2. Syncope in previous 3 months.
3. Unstable coronary artery disease.

   * Canadian Cardiovascular Society Class ≥ II angina.
   * Myocardial infarction in the past 3 months.
   * Symptomatic coronary artery disease with ≥50% stenosis on angiogram.
4. Moderate obstructive lung disease defined as forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) ratio < 0.7 and FEV1 < 70% predicted.
5. Active treatment for malignancy other than non-melanoma skin cancer in past 12 months.
6. Life expectancy < 12 months.
7. Actively listed for lung transplantation.
8. Cognitive, sensory, or musculoskeletal limitation that precludes participation in an exercise program, according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-03 (Estimated); Primary Completion 2022-11-03 (Estimated); Study Completion 2022-11-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the mobile application-based home exercise program | 12 weeks
  Feasibility will be defined as all of following:
  1. Recruitment of 20 patients in an 10 month period (2 per month),
  2. Consent ratio >30% (number who consent/number of eligible patients)
  3. Dropout rate < 20%
  4. Patient adherence to the exercise program >50%. Adherence will be expressed as average number of sessions completed per week over a 3-month period. A total adherence of >70% will be considered excellent, 50-70% will be considered acceptable

SECONDARY OUTCOMES:
Adverse events | 12 weeks
  Safety will be determined by patient-reported adverse events and serious adverse events.
Change in six-minute walking distance (6MWD) from baseline (relative and absolute). | Baseline, 12 weeks
  Measured according to American Thoracic Society guidelines for 6MWD
Change in maximal oxygen consumption (V'O2 peak) | Baseline, 12 weeks
  Measured by incremental symptom-limited cardiopulmonary exercise test.
Change in oxygen pulse (O2 pulse) | Baseline, 12 weeks
  Measured by incremental symptom-limited cardiopulmonary exercise test.
Change in ventilatory efficiency (V'E/V'CO2 slope and nadir) | Baseline, 12 weeks
  Measured by incremental symptom-limited cardiopulmonary exercise test.
Change in echocardiographic markers of right ventricular size and function. | Baseline, 12 weeks
  Measured with 2-dimensional and 3-dimensional transthoracic echocardiography
Change in EmPHasis-10 score from baseline. | Weekly for 12 weeks
  EmPHasis-10 is a simple 10-item disease-specific quality of life measurement. Scale 0-50. Higher EmPHasis-10 scores reflect worse quality of life.
Change in PRAISE self-efficacy score. | Weekly for 12 weeks
  Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) score is a validated self-efficacy score designed for the pulmonary rehabilitation population and is composed of 15 items. Each item is scored from 1 to 4 with a total range from 15 to 60. Higher scores indicate higher levels of self-efficacy.
Change in Living with Pulmonary Hypertension score from baseline. | Weekly for 12 weeks
  Living with Pulmonary Hypertension is a disease-specific quality of life score that is more widely validated than EmPHasis-10. Living with Pulmonary Hypertension questionnaire comprises 21 items and is responded to on a 6-point Likert scale ranging from 0 'No' to 5 'very much'. The total score ranges from 0 to 105. Higher scores indicate that the patients are more affected by their medical condition (worse quality of life).
Change in N-terminal-pro-brain natriuretic peptide (NT-proBNP) from baseline. | Weekly for 12 weeks
  NT-proBNP is a blood biomarker of right ventricular dysfunction.
Proportion of patients improving at ≥1 World Health Organization/New York Heart Association (WHO/NYHA) functional class. | Weekly for 12 weeks
  WHO/NYHA functional class is a subjective measure of functional capacity and symptoms.
Patient Satisfaction and Usability Questionnaire. | Weekly for 12 weeks
  This is a custom made questionnaire with qualitative open-ended questions and questions on a 5-point Likert scale from 1 (Very Dissatisfied) to 5 (Very Satisfied). Information will be used to refine the app and the exercise program for a subsequent trial.
Change in background step counts and/or actigraphy from baseline. | Baseline, 12 weeks
  This will serve to monitor study groups for baseline activity level as well as overall increased activity according to allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Weatherald, MD, Principal Investigator — University of Calgary
Locations (1):
- Peter Lougheed Centre (PLC), University of Calgary, Calgary, Alberta, Canada